CLINICAL TRIAL: NCT06957821
Title: Study to Image Inflammatory Activity of a Fluorescence Imaging Agent in Excised Human Artery Plaques
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024P002945; 5R01HL165453-03 (NIH)
Record Dates: First submitted 2025-05-02; First posted 2025-05-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Carotid Artery Diseases; Peripheral Arterial Disease
MeSH Terms: conditions — Carotid Artery Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEGULICIANINE (LUMISIGHT) (Experimental): Twenty (20) participants will receive 1.0 mg/kg of LUMISIGHT
  Interventions: Drug: Pegulicianine
- Normal Saline (Placebo Comparator): Five(5) participants will receive saline injections and be considered controls
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pegulicianine — Pegulicianine (LUMISIGHT) Inflammatory activity
  Other Names: LUMISIGHT
  Arms: PEGULICIANINE (LUMISIGHT)
Other: Placebo — Control group for the study
  Arms: Normal Saline

SUMMARY:
Active inflammation plays a key role in causing Coronary Artery Disease (CAD) and Peripheral Arterial Disease (PAD). Since inflammation is so important in how these diseases start, are diagnosed, and treated, being able to see it clearly in each patient could lead to more personalized and effective care - and may help prevent heart attacks. Right now, there's no imaging technology available to clearly see inflammation inside the coronary arteries.

The investigators hope to learn how an imaging drug; called LUMISIGHT (Pegulicianine) can help detect inflammation in blood vessels compared with saline. If the investigators find out that LUMISIGHT is active in humans, the investigators might be able to use it for detecting plaque risk in the future.

DETAILED DESCRIPTION:
Objective of this research is to find out if a new imaging drug called LUMISIGHT can show inflammation inside blood vessels for participants with severe coronary and peripheral arterial disease. This will allow us to obtain information about diseases that cause inflammation in the heart and blood vessels.

On the day of the procedure, at least 2 hours before the surgery, consented study participants will be injected with either the LUMISIGHT or saline. Following the injection, study participants will be monitored and observed for 30 minutes for any allergic reactions. Study participants will then undergo the standard of care surgery for their clinical care. During the procedure, surgeon will take out blocked pieces of subjects' blood vessel for clinical care. The investigators will get these discarded pieces and image it with a special imaging system developed by the Tearney Lab. This system uses a thin tube with a light-based camera (called Optical Coherence Tomography-Near Infra Red Fluorescence or OCT-NIRF) to capture detailed images.

ELIGIBILITY:
Inclusion Criteria:

* Must have an established diagnosis of severe carotid or peripheral arterial disease (ischemic or aneurysmal) requiring surgery and be sufficiently healthy to undergo surgery
* Must be age of 18 years or older
* Must be able to give informed consent
* Women with childbearing potential must have a negative pregnancy test
* Estimated glomerular filtration rate ≥ 60 mL/min/1.73 m2 (mild renal impairment

Exclusion Criteria:

* History of allergic reaction to oral or intravenous contrast agents
* History of allergic reaction to polyethylene glycol (PEG)
* History of allergic or anaphylactic reactions
* Participants who have taken an investigational drug within 14 days of enrollment.
* Participants with hemodynamic instability
* Any history of renal failure (estimated Glomerular Filtration Rate (eGFR) <60ml/min/1.73 m2)
* Pregnant or lactating females
* Participants with uncontrolled hypertension defined as persistent systolic blood pressure > 180 mm Hg, or diastolic blood pressure > 110 mm Hg; those subjects with known HTN should be under these values while under pharmaceutical therapy
* Severe concurrent illnesses including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, COPD or asthma requiring hospitalization within the past 12 months, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Demonstrate lumisight fluorescence activity in lumisight cohort vs controls | 2-6 hours
  Mean difference in plaque for fluorescence ratio to show that fluorescence in the Lumisight cohort is 2 fold greater than that of the control

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No